CLINICAL TRIAL: NCT03605862
Title: A Phase III, Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide in the Treatment of Colds Due to Enterovirus/Rhinovirus Infection
Brief Title: Efficacy and Safety of Nitazoxanide in the Treatment of Colds Due to Enterovirus/Rhinovirus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM08-3005
Record Dates: First submitted 2018-07-18; First posted 2018-07-30 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Enterovirus; Rhinovirus
Keywords: Enterovirus; Rhinovirus
MeSH Terms: conditions — Enterovirus Infections | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Active Comparator): Two Nitazoxanide 300 mg tablets orally twice daily for 5 days
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Two placebo tablets orally twice daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 600 mg administered orally twice daily for five days
  Other Names: NTZ (nitazoxanide); NT-300
  Arms: Nitazoxanide
Drug: Placebo — Placebo administered orally twice daily for five days
  Arms: Placebo

SUMMARY:
Trial to evaluate efficacy and safety of nitazoxanide in the treatment of colds due to Enterovirus/Rhinovirus infection

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind, placebo-controlled trial to evaluate efficacy and safety of nitazoxanide in the treatment of colds due to Enterovirus/Rhinovirus infection

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects at least 12 years of age
2. Presence of clinical signs and/or symptoms consistent with an acute illness compatible with EV/RV infection (each of the following is required):

   1. Presence of moderate or severe rhinorrhea defined as "attempting to relieve nasal symptoms by blowing, wiping, or sniffling at least twice per hour for any one hour within 12 hours preceding study entry," AND
   2. Presence of cough, sore throat or nasal obstruction.
3. Negative rapid influenza diagnostic test (required only if the subject has an oral temperature >100°F in the clinic or if the latest CDC weekly influenza report shows influenza prevalence "Regional" or higher for the institution's state). A result from a rapid influenza diagnostic test performed on the same day that informed consent is obtained will be sufficient to meet this criterion if documentation of test results is available as part of medical history.
4. Onset of illness no more than 40 hours before enrollment in the trial. Onset of illness is defined as the first time at which the subject experienced rhinorrhea, cough, sore throat or nasal obstruction.
5. Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the subject diary

Exclusion Criteria:

1. Persons requiring or anticipated to require in-hospital care
2. Cystic fibrosis
3. Cardiac arrhythmia
4. Immunologic disorders or receiving immunosuppressive therapy (e.g., for organ or bone marrow transplants, immunomodulatory therapies for certain autoimmune diseases)
5. Untreated HIV infection or treated HIV infection with a CD4 count below 350 cells/mm3 in the last 6 months
6. Persons with sickle cell anemia or other hemoglobinopathies
7. Poorly controlled insulin-dependent diabetes mellitus (HbA1C >8.0%)
8. Concurrent infection at the screening examination that requires systemic antimicrobial therapy
9. Females of childbearing potential who are either pregnant or sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an IUD, or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year - or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral oophorectomy.
10. Females who are breastfeeding
11. Receipt of any dose of NTZ within 30 days prior to screening
12. Prior treatment with any investigational drug therapy within 30 days prior to screening
13. Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies
14. Known sensitivity to NTZ or any of the excipients comprising the NTZ tablets
15. Subjects unable to take oral medications
16. Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol including completion of the subject diary

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1756 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossignol, M.D., Ph.D, Study Director — Romark Laboratories L.C.
Locations (41):
- United States (39):
  - Vanguard Study Site, Birmingham, Alabama
  - Vanguard Study Site, Pelham, Alabama
  - Vanguard Study Site, Hot Springs, Arkansas
  - Vanguard Study Site, Anaheim, California
  - Vanguard Study Site, Westminster, California
  - Vanguard Study Site, Wilmington, California
  - Vanguard Study Site, Miami, Florida
  - Vanguard Study Site, Orlando, Florida
  - Vanguard Study Site, Tampa, Florida
  - Vanguard Study Site, Stockbridge, Georgia
  - Vanguard Study Site, Blackfoot, Idaho
  - Vanguard Study Site, Meridian, Idaho
  - Vanguard Study Site, Nampa, Idaho
  - Vanguard Study Site, Evanston, Illinois
  - Vanguard Study Site, Valparaiso, Indiana
  - Vanguard Study Site, Louisville, Kentucky
  - Vanguard Study Site, New Orleans, Louisiana
  - Vanguard Study Site, Baltimore, Maryland
  - Vanguard Study Site, St Louis, Missouri
  - Vanguard Study Site, Missoula, Montana
  - Vanguard Study Site, Bellevue, Nebraska
  - Vanguard Study Site, Las Vegas, Nevada
  - Vanguard Study Site, Brooklyn, New York
  - Vanguard Study Site, Raleigh, North Carolina
  - Vanguard Study Site, Cincinnati, Ohio
  - Vanguard Study Site, Cleveland, Ohio
  - Vanguard Study Site, Columbus, Ohio
  - Vanguard Study Site, Dayton, Ohio
  - Vanguard Study Site, Medford, Oregon
  - Vanguard Study Site, East Providence, Rhode Island
  - Vanguard Study Site, Jackson, Tennessee
  - Vanguard Study Site, Milan, Tennessee
  - Vanguard Study Site, Austin, Texas
  - Vanguard Study Site, Carrollton, Texas
  - Vanguard Study Site, Houston, Texas
  - Vanguard Study Site, McAllen, Texas
  - Vanguard Study Site, Plano, Texas
  - Vanguard Study Site, Bountiful, Utah
  - Vanguard Study Site, St. George, Utah
- Puerto Rico (2):
  - Vanguard Study Site, Ponce
  - Vanguard Study Site, San Juan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitazoxanide | Placebo
Started | 872 | 884
Completed | 844 | 858
Not Completed | 28 | 26
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — "Other" reasons included failure to attend follow up visits or inability to use the eDiary. | 11 | 15

BASELINE CHARACTERISTICS:
Population: All subjects receiving at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide | Placebo | Total
Number analyzed (Participants) | 872 | 884 | 1756
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (14.82) | 37.3 (14.38) | 37.2 (14.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 613 | 567 | 1180
  Male | 259 | 317 | 576
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 173 | 175 | 348
  Hispanic | 124 | 150 | 274
  White | 551 | 536 | 1087
  Other | 24 | 23 | 47
Height [Mean (Standard Deviation); unit: cm] | 167.0 (9.83) | 168.3 (10.38) | 168.0 (10.11)
Weight [Mean (Standard Deviation); unit: kg] | 85.6 (25.03) | 85.8 (22.74) | 85.7 (23.90)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (8.05) | 30.3 (8.09) | 30.3 (8.07)
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 166 | 149 | 315
  Past Smoker | 120 | 123 | 243
  Never Smoked | 586 | 612 | 1198
Time from Onset of Symptoms at First Study Drug Intake (hours) [Mean (Standard Deviation); unit: hours] | 26.6 (9.1) | 26.3 (9.1) | 26.5 (9.1)
Respiratory Infection(s) [Count of Participants; unit: Participants]
  Adenovirus | 2 | 8 | 10
  Coronavirus (NL63, HKU1, 229E, or OC43) | 63 | 54 | 117
  Enterovirus/Rhinovirus | 286 | 298 | 584
  Human Metapneumovirus | 5 | 6 | 11
  Influenza A | 6 | 3 | 9
  Mycoplasma pneumoniae | 0 | 1 | 1
  Parainfluenza | 38 | 36 | 74
  Respiratory Syncytial Virus (RSV) | 19 | 18 | 37
Baseline Symptom Score, ITTI Population [Mean (Standard Deviation); unit: mean of patient-reported symptom ratings] — Subjects completed the FLU-PRO questionnaire during the Baseline visit. The questionnaire was scored according to the instrument algorithm (mean of symptom ratings with minimum possible score of 0 [symptoms absent] and maximum possible score of 4 [all symptoms very severe]). Population: Analysis population is the primary efficacy (intent-to-treat-infected, ITTI) population with laboratory-confirmed EV/RV infection.
  mean of patient-reported symptom ratings
    number analyzed (Participants) | 286 | 298 | 584
    (all) | 1.4 (0.59) | 1.4 (0.59) | 1.4 (0.59)
Baseline Patient-Reported Health Status, ITTI Population [Count of Participants; unit: Participants] — Subjects completed the inFLUenza Patient Reported Outcomes (FLU-PRO) questionnaire and global assessment questions during the Baseline visit. Baseline Health Status was assessed using the global assessment question, "Have you returned to your usual health?" with response options "yes" or "no". Population: Analysis population is the primary efficacy (intent-to-treat-infected, ITTI) population with laboratory-confirmed EV/RV infection.
  Participants
    At Usual Health: number analyzed (Participants) | 286 | 298 | 584
    At Usual Health | 35 | 42 | 77
    Not At Usual Health: number analyzed (Participants) | 286 | 298 | 584
    Not At Usual Health | 251 | 256 | 507
Baseline Illness Severity, ITTI Population [Count of Participants; unit: Participants] — Subjects completed the inFLUenza Patient Reported Outcomes (FLU-PRO) questionnaire and global assessment questions during the Baseline visit. Baseline Global Illness Severity was assessed using the global assessment question, "Overall, how severe were your cold symptoms today?" with response options "No cold symptoms today", "Mild", "Moderate", "Severe" or "Very Severe". Population: Analysis population is the primary efficacy (intent-to-treat-infected, ITTI) population with laboratory-confirmed EV/RV infection.
  Participants
    No cold symptoms: number analyzed (Participants) | 286 | 298 | 584
    No cold symptoms | 3 | 2 | 5
    Mild: number analyzed (Participants) | 286 | 298 | 584
    Mild | 40 | 34 | 74
    Moderate: number analyzed (Participants) | 286 | 298 | 584
    Moderate | 147 | 149 | 296
    Severe: number analyzed (Participants) | 286 | 298 | 584
    Severe | 83 | 93 | 176
    Very severe: number analyzed (Participants) | 286 | 298 | 584
    Very severe | 13 | 20 | 33
Baseline Symptom Interference in Activities, ITTI Population [Count of Participants; unit: Participants] — Subjects completed the inFLUenza Patient Reported Outcomes (FLU-PRO) questionnaire and global assessment questions during the Baseline visit. Baseline Symptom Interference in Activities was assessed using the question, "How much did your cold symptoms interfere with your usual activities today?" with response options "not at all", "a little bit", "somewhat", "quite a bit" or "very much". Population: Analysis population is the primary efficacy (intent-to-treat-infected, ITTI) population with laboratory-confirmed EV/RV infection.
  Participants
    Not at all: number analyzed (Participants) | 286 | 298 | 584
    Not at all | 48 | 37 | 85
    A little bit: number analyzed (Participants) | 286 | 298 | 584
    A little bit | 74 | 86 | 160
    Somewhat: number analyzed (Participants) | 286 | 298 | 584
    Somewhat | 87 | 94 | 181
    Quite a bit: number analyzed (Participants) | 286 | 298 | 584
    Quite a bit | 58 | 59 | 117
    Very much: number analyzed (Participants) | 286 | 298 | 584
    Very much | 19 | 22 | 41
Baseline Symptom Severity Compared to Yesterday, ITTI Population [Count of Participants; unit: Participants] — Subjects completed the FLU-PRO questionnaire and global assessment questions during the Baseline visit. Baseline Severity Compared to Yesterday was assessed using the question, "Overall, how were your cold symptoms today compared to yesterday?" with response options "much better", "somewhat better", "a little better", "about the same", "a little worse", "somewhat worse" or "much worse". Population: Analysis population is the primary efficacy (intent-to-treat-infected, ITTI) population with laboratory-confirmed EV/RV infection.
  Participants
    Much better than yesterday: number analyzed (Participants) | 286 | 298 | 584
    Much better than yesterday | 5 | 4 | 9
    Somewhat better than yesterday: number analyzed (Participants) | 286 | 298 | 584
    Somewhat better than yesterday | 11 | 10 | 21
    A little better than yesterday: number analyzed (Participants) | 286 | 298 | 584
    A little better than yesterday | 24 | 20 | 44
    About the same as yesterday: number analyzed (Participants) | 286 | 298 | 584
    About the same as yesterday | 89 | 80 | 169
    A little worse than yesterday: number analyzed (Participants) | 286 | 298 | 584
    A little worse than yesterday | 79 | 93 | 172
    Somewhat worse than yesterday: number analyzed (Participants) | 286 | 298 | 584
    Somewhat worse than yesterday | 47 | 48 | 95
    Much worse than yesterday: number analyzed (Participants) | 286 | 298 | 584
    Much worse than yesterday | 31 | 43 | 74

OUTCOME MEASURES:

1. Primary Outcome: Time From First Dose to Symptom Response Over 21 Days of Follow up Based Upon the FLU-PRO Instrument (Novel Endpoint)
Description: Subjects used the FLU-PRO questionnaire once daily in the evening to score the severity of 32 FLU-PRO symptoms. Symptom response was deemed achieved when the rating for each of the 32 FLU-PRO symptoms was ≤ its assigned threshold for 2 consecutive daily diary periods without use of symptom relief medication. The symptom response thresholds were developed by applying an algorithm to blinded symptoms data to select the set of 32 symptom thresholds most closely associated with patient-reported usual health.
Time Frame: Up to 21 days
Population: The primary efficacy (intent-to-treat infected, ITTI) population consisted of 584 subjects (N=286 in NTZ group, N=298 in Placebo group) with laboratory-confirmed Enterovirus/Rhinovirus (EV/RV) infection.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 286 | 298
hours | 122.5 [58 to 244] | 137.1 [75 to 243]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.4009, Gehan-Wilcoxon; Analysis was stratified by time from onset of symptoms, pre-enrollment symptom relief medication use, and presence of underlying lung conditions

2. Secondary Outcome: Time From First Dose to Ability to Perform All Normal Activities
Description: Subjects completed a diary including rating ability to perform normal activities on a scale from 0 (able to perform no normal activities) to 10 (able to perform all normal activities) daily in the evening. The time from first dose to ability to perform all normal activities is the time in hours between the first dose of study medication and that time when the subject first reported a score of "10" (able to perform all normal activities) for two consecutive daily diary periods without use of symptom relief medication.
Time Frame: Up to 21 days
Population: The efficacy (intent-to-treat infected, ITTI) population consisted of 584 subjects (N=286 in NTZ group, N=298 in Placebo group) with laboratory-confirmed Enterovirus/Rhinovirus (EV/RV) infection.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 286 | 298
hours | 174.3 [80 to 340] | 175.4 [105 to 318]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.1923, Gehan-Wilcoxon; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Proportions Experiencing Complications of EV/RV Infection
Description: Complications of colds due to EV/RV infection include pneumonia, otitis media, bronchitis, sinusitis, exacerbations of asthma or COPD, worsening of pre-existing health conditions, secondary infections requiring systemic antibiotic use, hospitalization due to cold or complications of the cold, and death due to cold or complications of the cold. Proportions experiencing complications of EV/RV infection were compared across treatment groups.
Time Frame: 28 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 286 | 298
Participants | 12 | 20
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.2057, Fisher Exact

4. Other Pre Specified Outcome: Time to Return to Usual Health
Description: Subjects completed the FLU-PRO questionnaire including global assessment questions daily in the evening. The time from first dose to ability to return to usual health is the time in hours from the first dose of study medication to the first time when the subject answered "Have you returned to your usual health?" with "yes" for two consecutive daily diary periods without the use of symptom relief medication.
Time Frame: 21 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 286 | 298
hours | 154.1 [80 to 320] | 174.9 [104 to 345]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.0712, Gehan-Wilcoxon; Analysis stratified by time from symptom onset at Baseline, pre-enrollment symptom relief medication use, and presence of underlying lung condition

5. Other Pre Specified Outcome: Proportion Positive for EV/RV by RT-PCR at Days 2, 3 and 7
Description: Proportion of subjects with nasopharyngeal swab collected testing positive for Enterovirus/Rhinovirus (EV/RV) infection by RT-PCR at each time point.
Time Frame: Days 2, 3, and 7
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 286 | 298
proportion of participants
  Day 2 | 0.81 | 0.81
  Day 3 | 0.79 | 0.79
  Day 7 | 0.66 | 0.76
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Comparison for study day 2; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Nitazoxanide vs Placebo; Comparison for study day 3; Test type: Superiority; p = 0.9142, Fisher Exact
Statistical Analysis 3: Comparison: Nitazoxanide vs Placebo; Comparison for study day 7; Test type: Superiority; p = 0.0132, Fisher Exact

6. Other Pre Specified Outcome: Analysis of Change From Baseline to Days 2, 3 and 7 in EV/RV Virus Titer
Description: Changes from baseline to day 2, baseline to day 3, and baseline to day 7 in EV/RV virus titer measured by quantitative RT-PCR. Samples negative for EV/RV were assigned the value of the limit of detection for the RT-PCR assay.
Time Frame: Days 2, 3, and 7
Population: Analysis population includes subjects with laboratory-confirmed EV/RV who were positive for EV/RV at the preceding swab collection time point. Per protocol, day 2 and 3 visits were optional.
Measure: Mean (Standard Error); unit: log10 RNA copies/mL
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 286 | 298
log10 RNA copies/mL
  Day 2: number analyzed (Participants) | 188 | 191
  Day 2 | -0.2203 (0.0934) | -0.4186 (0.0884)
  Day 3: number analyzed (Participants) | 175 | 174
  Day 3 | -0.5577 (0.1272) | -0.8282 (0.1053)
  Day 7: number analyzed (Participants) | 136 | 154
  Day 7 | -1.5113 (0.1373) | -1.6470 (0.1231)
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Comparison for day 2; Test type: Superiority; p = 0.1239, t-test, 2 sided
Statistical Analysis 2: Comparison: Nitazoxanide vs Placebo; Comparison for day 3; Test type: Superiority; p = 0.1022, t-test, 2 sided
Statistical Analysis 3: Comparison: Nitazoxanide vs Placebo; Comparison for day 7; Test type: Superiority; p = 0.46213, t-test, 2 sided

7. Other Pre Specified Outcome: Response Misclassification Rate Compared to Usual Health
Description: The proportion of patient diaries misclassified by the response definition used for the primary efficacy analysis compared to patient reported usual health. A diary was considered "misclassified" if the response definition predicted "responded" and the patient reported not being at usual health or if the response definition predicted "not responded" and the patient reported being at usual health.
Time Frame: 21 days
Population: The intent-to-treat-infected (ITTI) population consisted of all subjects positive for EV/RV at Baseline. Per the Statistical Analysis Plan, the response definition misclassification rate was to be calculated prior to unblinding including all data for subjects in the ITTI population.
Measure: Number; unit: n diaries misclassified/n diaries
Groups:
- ITTI Population: The intent-to-treat-infected (ITTI) population consisted of all subjects positive for EV/RV at Baseline.
Arm/Group | ITTI Population
Number analyzed (Participants) | 584
n diaries misclassified/n diaries | 0.21915

8. Post Hoc Outcome: Correlation Coefficient for Sustained Response and Return to Usual Health
Description: The correlation coefficient between sustained response and return to usual health was calculated for the pooled ITTI population (i.e., not by treatment group) as a measure of association between the primary endpoint response definition and its intended anchor, patient-reported return to usual health.
Time Frame: 21 days
Population: The intent-to-treat-infected (ITTI) population consisted of all subjects positive for EV/RV at Baseline. Consistent with calculation of the response definition misclassification rate, the correlation coefficient was calculated for all subjects in the ITTI population regardless of treatment group assignment.
Measure: Number; unit: correlation coefficient
Arm/Group | ITTI Population
Number analyzed (Participants) | 584
correlation coefficient | 0.43

9. Post Hoc Outcome: Time to Return to Usual Health, Modified ITTI Population
Description: Examination of Baseline disease characteristics revealed many subjects reporting via the Baseline FLU-PRO questionnaire that they are at their usual state of health, that symptoms do not interfere with any usual activities, and/or that symptoms are already improving. The pre-specified analysis of Time to Return for Usual Health was repeated for the population with Baseline subject-reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day. Time to Return to Usual Health is the time in hours between the first dose of study medication and the first time at which the subject answered "Have you returned to your Usual Health today?" via the daily FLU-PRO questionnaire with a "yes" for two consecutive diary periods without use of symptom relief medication.
Time Frame: 21 days
Population: Modified ITTI population consists of 387 subjects with laboratory-confirmed EV/RV infection and Baseline subject-reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day. Assessment was completed via the Baseline FLU-PRO questionnaire.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 183 | 204
hours | 153.7 [96 to 317] | 195.0 [123 to 365]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.0140, Gehan-Wilcoxon; Analysis stratified by time from symptom onset at first dose, pre-enrollment symptom relief medication use, and presence of underlying lung condition

10. Post Hoc Outcome: Time to Sustained Clinical Recovery
Description: Alternative means of endpoint construction were pursued to strengthen the relationship between symptoms-based endpoint measures and subject global assessments of health. Time to Sustained Clinical Recovery is an endpoint based on evidence of meaningful within-subject change sustained for the duration of the study. Time to Sustained Clinical Recovery is the time in hours from the first dose of study medication to the first time at which the subject reports a decrease in total FLU-PRO score from the previous diary with assessment that symptoms are at least "somewhat better than yesterday", no oral temperature ≥100.4 F in the prior 24 hours, and no future increase in any of the FLU-PRO domains except within validated background levels.
Time Frame: 21 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 286 | 298
hours | 171.4 [81 to 411] | 221.5 [103 to 504]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.0112, Gehan-Wilcoxon; Analysis stratified by time from onset at first dose, pre-enrollment symptom relief medication use, and presence of underlying lung condition

11. Post Hoc Outcome: Time to Sustained Clinical Recovery, Modified ITTI Population
Description: Analysis of Time to Sustained Clinical Recovery was repeated for the population with Baseline subject-reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day. Time to Sustained Clinical Recovery is the time in hours from the first dose of study medication to the first time at which the subject reports a decrease in total FLU-PRO score from the previous diary with assessment that symptoms are at least "somewhat better than yesterday", no oral temperature ≥100.4 F in the prior 24 hours, and no future increase in any of the FLU-PRO domains except within validated background levels.
Time Frame: 21 days
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 183 | 204
hours | 150.3 [81 to 322] | 244.1 [119 to 504]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p < 0.0001, Gehan-Wilcoxon; [statistical method as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: 28 days or until resolution of all adverse events, whichever occurred later.
Arm/Group | Nitazoxanide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/872 | 0/884
Serious Adverse Events (participants affected / at risk) | 4/872 | 1/884
Other Adverse Events (participants affected / at risk) | 200/872 | 58/884
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=872) | Placebo (N=884)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nitazoxanide (N=872) | Placebo (N=884)
Chromaturia (Renal and urinary disorders) | 153 | 10
Diarrhoea (Gastrointestinal disorders) | 53 | 38
Nausea (Gastrointestinal disorders) | 24 | 19

LIMITATIONS AND CAVEATS:
This study used a novel primary endpoint that was weakly correlated (r=0.43) with the anchor assessment of usual health, resulting in a primary analysis of questionable interpretability. The post-hoc analysis of Time to Sustained Recovery may be a more reliable endpoint given consistency with other endpoints (time to return to usual health, proportions experiencing complications, proportions positive for EV/RV).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT03605862/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03605862/SAP_001.pdf